CLINICAL TRIAL: NCT03760861
Title: First-in-man Trial of the Magnetic-controlled Balloon Inflation Mechanism of a Novel Ingestible Weightloss Microcapsule
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Collaborators: Nanyang Technological University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2018/00018
Record Dates: First submitted 2018-04-26; First posted 2018-11-30 (Actual); Last update posted 2018-12-17 (Actual); Status verified 2018-12

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: Open label pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Prototype Microcapsule Treatment Arm (Experimental): Intervention by placement of prototype weight-loss microcapsule in the stomach. Subjects will have a weight-loss microcapsule deployed endoscpically in the stomach. The intragastric balloon in the capsule will be inflated using an external magnet..
  Interventions: Device: Prototype Microcapsule Treatment

INTERVENTIONS:
Device: Prototype Microcapsule Treatment — The subject will be sedated and using an endoscope, a prototype microcapsule will be placed into the gastric corpus. Then, an external handheld magnet will be applied to inflate the balloon encapsulated in the microcapsule. Upon ascertaining the full inflation based on the endoscopic visualization, the investigator will wait another 10 minutes after that to observe how the subject feels before manually puncturing the balloon with needle knife, and retrieving the punctured balloon with the RothNet through the mouth.
  Other Names: Prototype weight-loss microcapsule placement in stomach

SUMMARY:
The objective of this study is to demonstrate the ease of deployment of a novel magnetically-controlled ingestible weight loss microcapsule* and the functionality of the magnetically controlled inflation of the balloon within the stomach.

DETAILED DESCRIPTION:
The objective of this study is to demonstrate the ease of deployment of a novel magnetically-controlled ingestible weight loss microcapsule and the functionality of the magnetically controlled inflation of the balloon within the stomach. Device comes in the form of a gelatine coated pill (Ø9.6mm x 27mm) . Once in the stomach, the device may be driven by external magnetic controllers which can control both its position and orientation. It allows flexible approach of the external magnetic fields in any axial directions of the device, and it also controls the inflation valve which controls the inflation of an attached balloon. The inflated balloon will partially fill up the stomach, giving the subject the feel of satiety to reduce his/her desire to eat more food.

ELIGIBILITY:
Inclusion Criteria

* Healthy subject, as evidenced by medical history
* Male or female aged 21-50 years of age
* Willing to undergo endoscopy to retrieve the balloon and to comply with all study procedures
* Ability to provide a signed and dated informed consent form

Exclusion Criteria:

* Individuals with anatomical abnormalities or functional disorders that may inhibit swallowing or passage through to the stomach
* Individuals with history or symptoms of clinically significant esophageal or gastric disorders, peptic ulcerations, hiatal hernia, patulous pyloric channel, erosive esophagitis, varices, angiectasia, Barrett's esophagus
* Individuals with bowel obstruction, congenital or acquired GI anomalies (e.g., atresias, stenosis, stricture, and/or diverticula), severe renal, hepatic, and/or pulmonary disease
* Individuals with bleeding disorders
* Individuals already having other bioenteric devices placed
* Individuals who have pace makers, metal implants or other devices on them
* Pregnant women
* Individuals unable to make/sign informed consent

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 3 (Estimated)
Dates: Start 2018-12-13 (Actual); Primary Completion 2019-12-01 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Successful inflation and maintenance of the fully inflated intragastric balloon. | 10 minutes
  A fully inflated intragastric balloon in the stomach that is maintained for at least 10 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Khek Yu Ho, MD, Principal Investigator — National University Health System
Locations (1):
- National University Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No